CLINICAL TRIAL: NCT06763926
Title: Intranasal Nafarelin Compared to Subcutaneous Triptorelin for Triggering Final Oocyte Maturation in Ovarian Stimulation: a Non-inferiority Randomised Controlled Clinical Trial
Brief Title: Intranasal Nafarelin For Triggering Oocyte Maturation
Acronym: INFORM
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion Dexeus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FSD-NAF-2024-11; 2024-516621-31-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-17; First posted 2025-01-08 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Fertility Disorders
Keywords: IVF; Infertility; Oocyte donor; GnRH agonist
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subcutaneous Triptorelin (Active Comparator): 200 mcg subcutaneous triptorelin 34-36 hours prior to planned oocyte collection
  Interventions: Drug: Subcutaneous Triptorelin
- Intranasal Nafarelin (Active Comparator): 800 mcg intranasal nafarelin 36 hours prior to planned oocyte collection
  Interventions: Drug: Intranasal nafarelin

INTERVENTIONS:
Drug: Subcutaneous Triptorelin — Oocyte donors will undergo progesterone-primed ovarian stimulation according to the standard operating protocol for the clinical unit. Specifically, on day 1 or 2 of the menstrual cycle, a transvaginal ultrasound will be performed to check the antral follicle count (AFC) and the absence of follicles >10mm. For participants taking oral contraceptives before the treatment, the pill-free interval before starting ovarian stimulation will be 5 days. Participants will administer exogenous gonadotropins (recombinant or urinary), along with 200mg oral micronized progesterone per day for pituitary suppression. Participants using any commercially available gonadotropin preparation will be eligible for inclusion.
  Once 3 follicles ≥18mm are observed, participants will be randomised to one of the study arms.
  In the control group, 200 mcg subcutaneous triptorelin will be administered 34-36 hours prior to planned oocyte collection.
  Arms: Subcutaneous Triptorelin
Drug: Intranasal nafarelin — Oocyte donors will undergo progesterone-primed ovarian stimulation according to the standard operating protocol for the clinical unit. Specifically, on day 1 or 2 of the menstrual cycle, a transvaginal ultrasound will be performed to check the antral follicle count (AFC) and the absence of follicles >10mm. For participants taking oral contraceptives before the treatment, the pill-free interval before starting ovarian stimulation will be 5 days. Participants will administer exogenous gonadotropins (recombinant or urinary), along with 200mg oral micronized progesterone per day for pituitary suppression. Participants using any commercially available gonadotropin preparation will be eligible for inclusion.
  Once 3 follicles ≥18mm are observed, participants will be randomised to one of the study arms.
  In the experimental group, 800 mcg intranasal nafarelin will be administered 34-36 hours prior to planned oocyte collection.
  Arms: Intranasal Nafarelin

SUMMARY:
This is a non-inferiority randomised, controlled clinical trial comparing subcutaneous triptorelin to intranasal nafarelin for the final maturation of oocytes in oocyte donors undergoing ovarian stimulation.

DETAILED DESCRIPTION:
Oocyte donors meeting the inclusion criteria will be randomised to receive triggering for final oocyte maturation with 200 micrograms of subcutaneous triptorelin (control group) or 800 micrograms of intranasal nafarelin (experimental group). The primary outcome is the number of mature (metaphase 2 (MII)) oocytes collected.

The study has been designed with a non-inferiority limit of a difference of 2 mature oocytes, with 80% power and one-sided alpha of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Oocyte donor
* Undergoing a progesterone-primed ovarian stimulation cycle (PPOS) with any commercially available gonadotropin preparation(s)
* BMI 18 - 30 kg/m2
* ≥10 follicles of ≥14mm average diameter on the last ultrasound prior to trigger administration
* Able and willing to provide written informed consent

Exclusion Criteria:

* Allergy or hypersensitivity to either of the study drugs
* Hypopituitarism
* Known pituitary tumour
* Contraindication to intranasal medication administration
* Previous poor response to agonist trigger

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Number of MII (metaphase 2) oocyte retrieved | Until study completion - average of 10-20 days

SECONDARY OUTCOMES:
Total number of oocytes retrieved | Until study completion - average of 10-20 days
Incidence of ovarian hyperstimulation syndrome | Until study completion - average of 10-20 days
Serum FSH levels 10-14 hours after trigger | 1 day after study medication
Serum LH levels at time of oocyte collection | 2 days after study medication
Serum FSH levels at time of oocyte collection | 2 days after study medication
Serum progesterone levels at time of oocyte collection | 2 days after study medication
Participant-reported pain | Until study completion - average of 10-20 days
  . Participant-reported pain (measured using a visual analogue scale from 0 (no pain) to 10 (severe pain))
Medication ease of use | Until study completion - average of 10-20 days
  Medication ease of use (measured using a visual analogue scale from 0 (very easy) to 10 (very difficult))
Medication preference | Until study completion - average of 10-20 days
  Medication preference (measured using a 5-point Likert scale from (a) "I would strongly prefer the nasal spray" to (e) "I would strongly prefer the injection")
Adverse events | Until study completion - average of 10-20 days

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos P Polyzos, MD, PhD, Principal Investigator — Dexeus Fertility
Locations (4):
- Spain (4):
  - Dexeus Mujer Sabadell, Sabadell, Barcelona
  - Dexeus Mujer Sant Cugat, Sant Cugat del Vallès, Barcelona
  - Dexeus Mujer Reus, Reus, Tarragona
  - Departamento de Ginecología Obstetricia y Reproducción. Hospital Universitari Dexeus, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Youssef MA, Van der Veen F, Al-Inany HG, Mochtar MH, Griesinger G, Nagi Mohesen M, Aboulfoutouh I, van Wely M. Gonadotropin-releasing hormone agonist versus HCG for oocyte triggering in antagonist-assisted reproductive technology. Cochrane Database Syst Rev. 2014 Oct 31;2014(10):CD008046. doi: 10.1002/14651858.CD008046.pub4. PMID 25358904
- [Background] V. Donno, A. R. Neves, S. Garcia Martinez, N. P. Polyzos. O-074 Dual trigger is not superior to GnRH Agonist alone for final oocyte maturation in elective fertility preservation. A Randomized Controlled Trial. Hum Reprod. 2024;39(Supp 1).
- [Background] Davenport MJ, MacLachlan VB, Vollenhoven BJ, Talmor AJ, Healey M. How we trigger matters: intranasal GnRH-agonist trigger may reduce oocyte maturation compared to subcutaneous administration in ICSI cycles. Fertility and Sterility. 2019
- [Background] Bar Hava I, Yafee H, Omer Y, Humaidan P, Ganer Herman H. GnRHa for trigger and luteal phase support in natural cycle frozen embryo transfer - A proof of concept study. Reprod Biol. 2020 Sep;20(3):282-287. doi: 10.1016/j.repbio.2020.07.009. Epub 2020 Jul 30. PMID 32741721
- [Background] Bar-Hava I, Mizrachi Y, Karfunkel-Doron D, Omer Y, Sheena L, Carmon N, Ben-David G. Intranasal gonadotropin-releasing hormone agonist (GnRHa) for luteal-phase support following GnRHa triggering, a novel approach to avoid ovarian hyperstimulation syndrome in high responders. Fertil Steril. 2016 Aug;106(2):330-3. doi: 10.1016/j.fertnstert.2016.04.004. Epub 2016 Apr 22. PMID 27114332
- [Background] Golan A, Weissman A. Symposium: Update on prediction and management of OHSS. A modern classification of OHSS. Reprod Biomed Online. 2009 Jul;19(1):28-32. doi: 10.1016/s1472-6483(10)60042-9. PMID 19573287
- See also: Related Info — http://www.dexeus.com